CLINICAL TRIAL: NCT00982410
Title: Managing Chronic Pain in Veterans With Substance Use Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAC 09-047
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Pain
Keywords: pain; alcohol; illicit drugs; pain management
MeSH Terms: conditions — Chronic Pain; Pain; Substance-Related Disorders; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): cognitive-behavioral treatment (CBT) interventions to manage pain and decrease substance use abuse/misuse
  Interventions: Behavioral: cognitive-behavioral treatment
- Arm 2 (Placebo Comparator): educational supportive group
  Interventions: Behavioral: educational supportive group

INTERVENTIONS:
Behavioral: cognitive-behavioral treatment — cognitive-behavioral treatment (CBT) interventions to manage pain and decrease substance use abuse/misuse
  Arms: Arm 1
Behavioral: educational supportive group — A control condition providing social support and education about pain and/or drug use.
  Arms: Arm 2

SUMMARY:
The proposed project will provide crucial data on the effectiveness of a pain management intervention designed for veterans with co-occurring pain and substance use disorders. The development of an empirically validated psychosocial intervention for managing pain and substance misuse could greatly enhance the current set of options for treating this large and understudied group of veterans.

DETAILED DESCRIPTION:
Background: Chronic non-cancer pain and substance use disorders frequently co-occur in VA primary care and addictions treatment settings. The treatment for pain is complicated in veterans with a history of alcohol or drug misuse because of a potential for abuse and diversion of many prescription pain medications. Thus, treatment providers are left without successful and empirically-supported methods for treating the large number of patients with chronic pain who also have past or current substance use disorders. One potential strategy is to use cognitive-behavioral treatment (CBT) interventions to manage pain and decrease substance use abuse/misuse. Psychosocial interventions such as CBT have demonstrated efficacy for reducing pain and improving functioning in persons with a broad spectrum of pain-related problems. However, this form of treatment has not been explicitly tested in patients with co-occurring substance use disorders. Determining the effectiveness of a psychosocial intervention targeting both pain and substance use disorders would greatly increase the available treatment options for veterans with these conditions.

Project Objectives: This project is designed to test the effect of a CBT intervention for patients with chronic pain who are already engaged in VA treatment for substance use disorders compared to an educational supportive condition on measures of pain intensity, pain-related disability and pain-tolerance. A set of secondary analyses will examine if group CBT compared to the educational supportive condition is associated with greater reductions in illicit substance use over the follow-up time period and whether during-treatment reductions in pain mediate the effect of treatment assignment on later substance use. Finally, a series of secondary analyses will explore whether the hypothesized mechanisms of action for the CBT intervention mediate the effect of this intervention on pain intensity and pain tolerance.

Methods: The proposed study is a randomized controlled trial of group-based CBT compared to an educational supportive condition in patients currently receiving drug and alcohol treatment. At least 128 Veterans with alcohol or drug abuse or dependence and at least moderate pain currently treated in the Ann Arbor VA Substance Use Disorder treatment clinic will be assessed at baseline and then randomly assigned to one of these two conditions. These patients will be re-assessed at 3-months (i.e. immediately post treatment), 6-months and 12-months. The primary outcomes will be pain intensity, pain-related disability and pain tolerance. Mixed model regression analyses will be used for all primary analyses to estimate between-group differences in changes in individual slopes over time. Finally, a series of secondary analyses will explore (a) whether the intervention influences post-treatment substance use, (b) if change in pain during treatment mediates the effect of the intervention on subsequent substance use and (c) whether the hypothesized mechanisms of action for the CBT intervention mediate the effect of this intervention on pain intensity and pain tolerance.

ELIGIBILITY:
Inclusion Criteria:

* A report of pain of at least moderate or greater over the three months prior to baseline assessment as indicated by an average score of four or greater on the Numeric Rating Scale of pain intensity (NRS-I; Farrar et al. 2001);
* Completion of an intake assessment in the Ann Arbor VA's SUD clinic within the three months prior to baseline assessment. The pain-related inclusion criterion will be used to ensure that participants are experiencing elevated levels of pain and, consequently, are appropriate for pain-related treatment.

Exclusion Criteria:

* Acute suicidality based on responses on the Beck Depression Inventory (BDI) confirmed by in-depth assessment of patient by the research associate;
* Psychiatric condition that precludes participation in outpatient group treatment based on:

  * a Mini-Mental State Examination (MMSE; Folstein et al. 1975) score less than 21,
  * psychiatric hospitalization within the past month, or
  * endorsement of current psychotic symptoms on the Brief Symptom Inventory (BSI; Derogatis 1993) combined with noticeable bizarre thoughts or behavior during the interview;
* Inability to speak and understand English; and
* The inability to give informed, voluntary, written consent.

Decisions about exclusion criteria 1 and 2 will be made using a combination of self-reported symptoms and researcher's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Ilgen, PhD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Behavioral Treatment Group (CBT): An intervention treatment group to manage pain and decrease substance use abuse/misuse
  Cognitive-behavioral treatment (CBT) interventions to manage pain and decrease substance use abuse/misuse
  Each condition consisted of 10 weekly sessions, lasting approximately one hour in length, led by masters level therapists (i.e., social workers) at the Ann Arbor Veterans Affairs Medical Center (VAMC). Participants continued to receive their standard of care at the VA. The CBT condition's main foci included cognitive skills, acceptance skills, behavioral skills, life skills and concepts, and relaxation exercises.
- Educational Supportive Group: A control condition providing social support and education about pain and/or drug use.
  Each condition consisted of 10 weekly sessions, lasting approximately one hour in length, led by masters level therapists (i.e., social workers) at the Ann Arbor VAMC. Participants continued to receive their standard of care at the VA. The Educational Supportive Group condition's provided psycho-education about topics such as substance abuse, chronic pain, and how to maintain a healthy lifestyle
Period: 3-month Follow-up Assessment
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Started | 65 | 66
Completed | 56 | 53
Not Completed | 9 | 13
Not completed — Could not reach to schedule | 8 | 9
Not completed — Scheduled, no-show | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: 6-month Follow-up Assessment
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Started | 65 (n=65 : intent to treat. Some persons missed follow-up assessment without withdrawing from study.) | 64 (n=2 persons withdrew before 3-mo. f/u, reducing pool of participants to N=64 with intent to treat.)
Completed | 59 | 53
Not Completed | 6 | 11
Not completed — Could not reach to schedule | 5 | 7
Not completed — participant no transportation | 1 | 0
Not completed — incarceration | 0 | 2
Not completed — patent surgery | 0 | 1
Not completed — scheduled, no-show | 0 | 1
Period: 12-month Follow-up Assessment
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Started | 65 (n=65 : intent to treat. Some persons missed follow-up assessment without withdrawing from study.) | 64 (n=2 persons withdrew before 3-mo. f/u, reducing pool of participants to N=64 with intent to treat.)
Completed | 56 | 55
Not Completed | 9 | 9
Not completed — Death | 0 | 2
Not completed — could not reach to schedule | 6 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — incarceration | 2 | 1
Not completed — scheduled, no-show | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cognitive Behavioral Treatment Group: An intervention treatment group to manage pain and decrease substance use abuse/misuse
  Cognitive-behavioral treatment (CBT) interventions to manage pain and decrease substance use abuse/misuse
  Each condition consisted of 10 weekly sessions, lasting approximately one hour in length, led by masters level therapists (i.e., social workers) at the Ann Arbor VAMC. Participants continued to receive their standard of care at the VA. The CBT condition's main foci included cognitive skills, acceptance skills, behavioral skills, life skills and concepts, and relaxation exercises.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Treatment Group | Educational Supportive Group | Total
Number analyzed (Participants) | 65 | 66 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 64 | 128
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.2) | 51.3 (10.1) | 51.5 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 58 | 58 | 116
Self-reported average pain level in the past week via NRS-1 [Mean (Standard Deviation); unit: units on a scale] — Rate your pain, on average over the past week. Scale ranging from 0 (no pain) to 10 (worst possible pain). Average pain within last week.
  units on a scale | 7.15 (1.61) | 7.09 (1.62) | 7.14 (1.62)
WHY-MPI: Pain Severity Score [Mean (Standard Deviation); unit: units on a scale] — To measure pain-severity, we will use the Interference subscale of the West Haven-Yale Multidimensional Pain Inventory (WHYMPI). The WHYMPI/MPI is designed to be a brief, psychometrically-valid, and comprehensive assessment of the chronic pain experience for an individual. The WHY-MPI scores range from 0 to 6 with lower scores representing a better outcome.
  units on a scale | 4.31 (0.97) | 4.31 (0.89) | 4.31 (0.94)
WHY-MPI General Activity [Mean (Standard Deviation); unit: units on a scale] — West Haven-Yale M Pain Inventory: Score is a composite construct designed to assess the extent to which physical pain impacts daily living. Aspects include ability to perform chores inside home, activities away from home, and social functioning. WHY-MPI General Activity Score ranges from 0-6; high scores represent better outcomes.
  units on a scale | 2.24 (0.82) | 2.04 (0.89) | 2.14 (0.86)
CPSS: Self- efficacy for physical functioning (FSE score) [Mean (Standard Deviation); unit: units on a scale] — The CPSS is a 22-item questionnaire designed to measure chronic pain patients' perceived self-efficacy to cope with the consequences of chronic pain (Anderson et al. 1995). The CPSS has three primary subscales: self-efficacy for pain management (PSE), self-efficacy for physical function (FSE) and self-efficacy for coping with symptoms (CSE). These scales have high reliability. Scores range from 10-100, with higher scores representing a better outcome.
  units on a scale | 63.9 (22.0) | 60.6 (21.9) | 62.3 (21.9)
CPSS: self-efficacy for pain management (PSE score) [Mean (Standard Deviation); unit: units on a scale] — The CPSS is a 22-item questionnaire designed to measure chronic pain patients' perceived self-efficacy to cope with the consequences of chronic pain (Anderson et al. 1995). The CPSS has three primary subscales: self-efficacy for pain management (PSE), self-efficacy for physical function (FSE) and self-efficacy for coping with symptoms (CSE). These scales have high reliability. Scores range from 10-100, with higher scores representing a better outcome.
  units on a scale | 50.2 (22.1) | 42.1 (19.8) | 46.3 (21.3)
Alcohol abuse or alcohol dependence [Number; unit: participants] — University of Arkansas Substance Abuse Outcomes Module (SAOM; Smith et al. 1996). 25-item self-report measure designed to assess the severity of alcohol and drug problems (coefficient alpha = .9). Persons classified as alcohol abusers (a) had no dependence, but (b) did meet the criteria for abuse. Alcohol use questions concern the number of days of alcohol use, the average consumption per drinking day, the maximum consumption, and the number of binge days (more than five drinks consumed). Standard drinks are explained prior to asking these questions.
  participants
    Abuse or Dependence | 38 | 35 | 73
    No Abuse; No Dependence | 27 | 31 | 58
Drug abuse or drug dependence [Number; unit: participants] — University of Arkansas Substance Abuse Outcomes Module (SAOM; Smith et al. 1996). 25-item self-report measure designed to assess the severity of alcohol and drug problems. Persons classified as drug abusers (a) had no dependence, but (b) did meet the criteria for abuse on one or more substance. If a person met criteria for abuse on one substance and dependence on another, they were classified as drug-dependent. Persons with no abuse and no dependence did not meet criteria for abuse or dependence. Based on use of cannabis, cocaine, opioids, or stimulants in past 4 weeks.
  participants
    Any drug abuse or dependence | 30 | 33 | 63
    No Abuse; No dependence | 35 | 33 | 68
Prescription opioid misuse [Number; unit: participants] — Binary variable; based on 4 COMM (17-item self-report measure of current aberrant drug-related behavior over the past 30 days and answer choices range from 0 (never) to 4 (often)), questions pertaining to a) taking more Rx opioids than prescribed, b) taking Rx opioids prescribed to someone else, c) borrowing Rx opioids from someone else, and d) using Rx opioids for non-pain symptoms. Persons reporting any history of doing any of these 4 things were classified into opioid misuse categories, and persons who answered "never" to all 4 questions were classified as not misusing opioids.
  participants
    Ever misused Rx opioids | 37 | 39 | 76
    Never misused Rx opioids | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity, as Measured by Average Pain Within the Last Week (NRS-1)
Description: The outcome measure below represents the average pain levels in each Arm/Group, across the entire follow-up period. Average pain in the last week (NRS-1) is a scale ranging from 0 (no pain) to 10 (worst possible pain). The results reported below are based on longitudinal repeated measures modeling, adjusted for baseline NRS-1 average pain level. The variance was modeled to account for time interval (3-mo, 6-mo, 12-mo), and for session block; at the time of randomization, participants were assigned to blocks for a series of 10 sessions, in parallel for the intervention and control. Session blocks were utilized as a blocking variable to address between-block variation.
Time Frame: Baseline, 3-, 6-, & 12-months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Treatment Group | Educational Supportive Group
Number analyzed (Participants) | 65 | 64
units on a scale | 5.82 (0.24) | 6.47 (0.18)
Statistical Analysis 1: Comparison: Cognitive Behavioral Treatment Group vs Educational Supportive Group; Ho: There was no difference in average pain level across the follow-up period, between CBT group and Educational support group; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Adjusted for baseline NRS-1 pain level. Time interval and therapy session block were utilized to model the variance; Mean Difference (Final Values) = -0.6489, 95% CI 2-sided [-1.2255 to -0.07220], Standard Error of Mean 0.29 — EUC (Arm 2) was referent. Estimation parameter = value for Cognitive Behavior Treatment group minus value for Educational Support group

2. Primary Outcome: The Impact of Pain on Activities and Functioning: General Activity Score (WHY MPI)
Description: The WHY MPI General Activity score is a composite construct designed to assess the extent to which physical pain impacts various aspects of daily living. Aspects include ability to perform chores inside the home, activities away from the home, and social functioning. The outcome measure below represents the average pain levels in each Arm/Group, across the entire follow-up period, and was adjusted for baseline WHY MPI General Activity score.
Time Frame: Baseline, 3-,6-, 12-month
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Cognitive Behavioral Treatment Group (CBT): An intervention treatment group to manage pain and decrease substance use abuse/misuse
  Cognitive-behavioral treatment (CBT) interventions to manage pain and decrease substance use abuse/misuse
  Each condition consisted of 10 weekly sessions, lasting approximately one hour in length, led by masters level therapists (i.e., social workers) at the Ann Arbor VAMC. Participants continued to receive their standard of care at the VA. The CBT condition's main foci included cognitive skills, acceptance skills, behavioral skills, life skills and concepts, and relaxation exercises.
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 65 | 64
units on a scale | 2.24 (0.08) | 2.00 (0.06)
Statistical Analysis 1: Comparison: Cognitive Behavioral Treatment Group (CBT) vs Educational Supportive Group; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Adjusted for baseline WHY MPI General Activity score. Time interval and therapy session block were utilized to model the variance; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.034 to 0.466] — Education Support group was referent. Mean difference = value for CBT group minus value for Educational Support group

3. Primary Outcome: Alcohol Use
Description: #days used alcohol in the past 30 days, as assessed via timeline follow-back(TLFB) calendars. #days in a controlled environment (e.g. hospitalization, incarceration) also recorded to identify the duration of days at risk. The outcome measure below represents the average #days alcohol use in each Arm/Group, across the entire follow-up period, and was adjusted for baseline TLFB #days used alcohol.
Time Frame: Baseline, 3-, 6-, 12- months
Measure: Mean (Standard Error); unit: #Days used
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 65 | 64
#Days used | 2.05 (0.58) | 4.04 (0.92)
Statistical Analysis 1: Comparison: Cognitive Behavioral Treatment Group (CBT) vs Educational Supportive Group; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Adjusted for baseline #days of alcohol use. Time interval and therapy session block were utilized to model the variance

4. Primary Outcome: Drug Use
Description: # days used illicit drugs in the past 30 days, as assessed via timeline follow-back (TLFB) calendars. Use of illicit drugs and misuse of prescription drugs (e.g., Rx opioids) were recorded for the 30 days prior to the follow-up visit. #days in a controlled environment (e.g., hospitalization, incarceration) also recorded to identify the duration of days at risk. The outcome measure below represents the average #days drug use in each Arm/Group, across the entire follow-up period, and was adjusted for baseline TLFB #days used illicit drugs.
Time Frame: Baseline, 3-, 6-, 12- months
Measure: Mean (Standard Error); unit: #Days used
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 65 | 64
#Days used | 6.82 (1.72) | 6.85 (1.75)
Statistical Analysis 1: Comparison: Cognitive Behavioral Treatment Group (CBT) vs Educational Supportive Group; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Adjusted for baseline #days illicit drug use. Time interval and therapy session block were utilized to model the variance. EUC group was referent

5. Primary Outcome: Pain Tolerance
Description: Pain tolerance was measured by the amount of time the participant could hold their hand immersed in a vessel of cold water in seconds. The maximum allowed duration of the test was two minutes. The outcome measure below represents the average duration of task in each Arm/Group, across the entire follow-up period, and was adjusted for baseline level of pain tolerance.
Time Frame: Baseline, 3-,6-,12-months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 65 | 64
seconds | 70.2 (3.2) | 65.5 (3.8)
Statistical Analysis 1: Comparison: Cognitive Behavioral Treatment Group (CBT) vs Educational Supportive Group; Test type: Superiority or Other; p > 0.05, Mixed Models Analysis; Adjusted for baseline pain tolerance. Time interval and therapy session block were utilized to model the variance; Mean Difference (Final Values) = 4.66, 95% CI 2-sided [-5.00 to 14.32] — Educational Support group = referent. Estimation parameter = CBT group minus EUC group, adjusted for BL pain tolerance. Cold tolerance distribution had ceiling and floor effects; and, ~20% of participants refused cold tolerance task in follow-up

6. Secondary Outcome: Self-efficacy of Pain Management
Description: As measured via CPSS PSE score at each time point. The CPSS is a 22-item questionnaire designed to measure chronic pain patients' perceived self-efficacy to cope with the consequences of chronic pain (Anderson et al. 1995). The CPSS PSE subscale is a measure of self-efficacy for pain management. These scales have high reliability. Scores range from 10-100, with higher scores representing a better outcome. The outcome measure below represents the average CPSS PSE score in each Arm/Group, across the entire follow-up period, and was adjusted for baseline CPSS PSE.
Time Frame: Baseline, 3-, 6-, 12- months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 65 | 64
units on a scale | 57.9 (2.15) | 47.59 (2.40)
Statistical Analysis 1: Comparison: Cognitive Behavioral Treatment Group (CBT) vs Educational Supportive Group; Test type: Superiority or Other; p < 0.005, Mixed Models Analysis; Adjusted for baseline CPSS PSE score. Time interval and therapy session block were utilized to model the variance. EUC group was referent; Mean Difference (Final Values) = 10.28, 95% CI 2-sided [3.93 to 16.63] — Adjusted for baseline CPSS PSE score. EUC group was referent. Mean difference = value for CBT minus value for Educational Support group

7. Secondary Outcome: Self-efficacy of Physical Functioning
Description: The CPSS is a 22-item questionnaire designed to measure chronic pain patients' perceived self-efficacy to cope with the consequences of chronic pain (Anderson et al. 1995). The CPSS subscale, self-efficacy for physical function (FSE), utilized to assess management of pain-related disability, with respect to several aspects of daily functioning. This scale have high reliability. Scores range from 10-100, with higher scores representing a better outcome. The outcome measure below represents the average CPSS FSE score in each Arm/Group, across the entire follow-up period, and was adjusted for baseline level of CPSS FSE.
Time Frame: Baseline, 3-, 6-, 12- months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 65 | 64
units on a scale | 69.12 (2.01) | 61.57 (2.41)

8. Secondary Outcome: As-treated Analysis: Pain Intensity, as Measured by Average Pain Within the Last Week (NRS-1)
Description: Per study protocol, participants were asked to attend 10 sessions, which comprised the intervention for CBT participants and educational support for EUC participants. Some participants in each group did not attend any sessions, yet participated in follow-up assessments. The As-treated analysis was undertaken to evaluate the impact of the intervention, among participants that attended at least 1 session. As in the Primary Analysis, average pain last week (NRS-1) is a scale ranging from 0 (no pain) to 10 (worst possible pain). The results reported below are based on longitudinal repeated measures modeling, adjusted for baseline NRS-1 average pain level. The variance was modeled to account for time interval (3-mo, 6-mo, 12-mo), and for session block; at the time of randomization, participants were assigned to blocks for a series of 10 sessions, in parallel for the intervention and control. Session blocks were utilized as a blocking variable to address between-block variation
Time Frame: Baseline, 3-, 6-, 12-months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 55 | 47
units on a scale | 5.84 (0.21) | 6.47 (0.19)

9. Secondary Outcome: As-treated Analysis: The Impact of Pain on Activities and Functioning: General Activity Score (WHY MPI)
Description: The WHY MPI General Activity score is a composite construct designed to assess the extent to which physical pain impacts various aspects of daily living. The outcome measure below represents the average WHY MPI General Activity score in each Arm/Group, across the entire follow-up period, adjusted for baseline WHY MPI General Activity score, but restricted here to study participants that partook in at least one treatment group session.
Time Frame: Baseline, 3mo, 6mo, 12mo follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Cognitive Behavioral Treatment Group (CBT) | Educational Supportive Group
Number analyzed (Participants) | 55 | 47
units on a scale | 2.22 (0.08) | 1.95 (0.08)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Cognitive Behavioral Treatment Group | Educational Supportive Group
Serious Adverse Events (participants affected / at risk) | 0/65 | 3/66
Other Adverse Events (participants affected / at risk) | 0/65 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Treatment Group (N=65) | Educational Supportive Group (N=66)
Participant Death (General disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes